CLINICAL TRIAL: NCT04457635
Title: Effect of a 'Rapid-Return-to-work Program' in Mild Mental Disorders. A Randomized Controlled Trial.
Brief Title: Effect of a 'Rapid-Return-to-work Program' in Mild Mental Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Responsible Party: Principal Investigator, Aage Indahl, professor emeritus, The Hospital of Vestfold
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HVestfold
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Mental Disorder
Keywords: Return to Work; Brief Intervention
MeSH Terms: conditions — Mental Disorders | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor of primary outcome (sickness benefit) is masked for intervention allocation. Other outcome measures are assessed by patient questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief psychotherapy (brief PsT) (Experimental): The focus was on normalizing, accepting and coping with their present mental health complaints and their hindrance for work participation. Primarily, there was no intention to process previous pathogenic experiences. The standard duration was set on six sessions.
  Interventions: Behavioral: Psychotherapy
- Short psychotherapy (short-PsT) (Active Comparator): With more extended focus, there was besides coping of mental health and challenges concerning WP, an emphasis on both an extensive anamnesis and possibility to establish a so-called central theme based on previous or current challenging issues such as trauma, difficult childhood conditions, and personality-related issues. Additional aims of the intervention could include reducing symptoms and problematic behaviour and an improvement of home situation, with deeper focus on cognitive maladaptive coping strategies or dynamic repetitions. The number of sessions was aimed to be 20 on average
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy

SUMMARY:
This study is a pragmatic randomized controlled trial (RCT) evaluating the effect of brief versus short psychotherapy in subjects with substantial mental complaints.

DETAILED DESCRIPTION:
Running evaluations of the brief intervention (BI) at our outpatient clinic preceding to this study had given us the impression that the patients obtained a more active coping style towards their health problems with consequential enhanced work participation (WP). These evaluations, in addition to our experiences in BI for low back pain (LBP) has generated the current hypothesis of this study towards WP. Yet, the sustainability of WP and long-term effects on mental health remained questionable. In this pragmatic RCT the objective was to compare brief psychotherapy with focus on normalization and coping (Brief-PsT) with short-term psychotherapy of standard duration with more extended focus (Short-PsT), as otherwise used at the Mental Health services. The primary aim of this study was to assess differences in effect on WP and the secondary aim was to assess differences in clinical response. The investigators hypothesized that in the short term, Brief-PsT could facilitate or sustain WP in a superior fashion to Short-PsT in persons who are on, or at risk of sick leave due to mental health problems. Although the investigators expected a substantial long-term rate of clinical recovery and reduction in mental health-related symptoms in both groups, the investigators had no specific hypothesis regarding the extent and direction of possible group differences in these clinical measurements.

ELIGIBILITY:
Inclusion Criteria:

* 'mental complaints' was the main reason for referral to the outpatient clinic
* employed and on or at risk of sick leave

Exclusion Criteria:

* acute or severe pathology that required greater input than the clinic could offer,
* Sick-leave had > 9 months during the preceding 2 years

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in Return to Work (RTW) to 3 months follow-up | baseline - 3 months
  Transitions from baseline to 3 months follow-up in Work Participation degree
Change in Return to Work (RTW) to 1 year follow-up | baseline - 1 year
  Transitions from baseline to 1 year follow-up in Work Participation degree
Change in Return to Work (RTW) to 2 year follow-up | baseline - 2 year
  Transitions from baseline to 2 year follow-up in Work Participation degree

SECONDARY OUTCOMES:
Clinical recovery | 2 years
  A minimal score on both Beck Inventories (BDI ≤ 13 and BAI ≤ 9)

OTHER OUTCOMES:
Beck Depression Index - II (BDI) | baseline, 2 year follow-up
  Score 0-63, higher scores mean worse outcome
Beck Anxiety Index (BAI) | baseline, 2 year follow-up
  Score 0-63, higher scores mean worse outcome
Hopkins Symptoms Checklist-10 | baseline, 2 year follow-up
  Score 1-4, higher scores mean worse outcome
Subjective health complaints (SHC) | baseline, 2 year follow-up
  Score 0-29, higher scores mean worse outcome
Self-efficacy (GSES) | baseline - 2 year follow-up
  Score 1-4 , lower scores means worse outcome
Lfe satisfaction (LISAT) | baseline - 2 year follow-up
  Score 1-6, lower scores means worse outcome
Illness perception (bIPC) | baseline - 2 year follow-up
  Score 1-10, higher scores mean worse outcome
Fear avoidance beliefs -work (FABQ-work) | baseline - 2 year follow-up
  Score 0-7, higher scores mean worse outcome
Global Perceived Effect | 2 year follow-up
  Score 0-7, lower scores means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Aage Indahl, Prof.Dr, Study Director — Vestfol Hospital Trust

IPD SHARING:
Plan to Share IPD: No